CLINICAL TRIAL: NCT02682875
Title: The Evaluation With Artificial Neural Network of Pain Scales in Children
Brief Title: The Evaluation With Artificial Neural Network of Pain Scales in Children (ANN)
Acronym: ANN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra, Medical Doctor, Cukurova University
Other Study IDs: Zehra123
Record Dates: First submitted 2016-01-27; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The study evaluates with Artificial Neural Network (ANN) of pain scales in children. Pain of these patients' will be evaluated by many pain scales in the postoperative period.

DETAILED DESCRIPTION:
Pain of these patients' will be evaluated by many pain scales in the postoperative period. These scales include OUCHER, Visiuel Analog Scale, FLACC, Faces Pain Scale revise, Wong Baker Faces Scale, Faces Pain Scale, Numeric rating Scale, Verbal Rating Scale, CHEOPS and also age, blood pressure, respiratuar rate, heart rate will be recorded.

In the first step of this study, the parameters taken into account on widely used each pain scale practically and importance level of each parameter will be examined. The parameters taken into account in determining the degree of pain and degree of each pain scale will be recorded. Independent t-test of the pain scales will be analyzed whether different statistically. Pain scales used in the application at conclusion statistical analysis will be grouped.

In addition, parameters considered to be effective on pain (pulse, blood pressure, etc.) will be determined and also recorded. The degree of importance on pain of the current scales and other parameters to be determined and as result, new pain scale will be created. While determining the the level of importance will be utilized from the analytic hierarchy process (AHP). Making binary comparisons between AHP and parameters, the level of importance and weightiness score of each parameter will be determined. The mathematical formulation of the pain points will be presented considering AHP weightiness score of each parameter.

Although pain scores obtained mathematically, pain score with Artificial Neural Network (ANN) will be estimated considering the parameters that impact on the pain score.

The final step, the creation of new pain scale comparing the pain scores obtained by mathematical formulation and Artificial Neural Network and, it is intended to be compared with the current scales.

ELIGIBILITY:
Inclusion Criteria:

* 2 months -18 years
* Children undergoing elective surgery

Exclusion Criteria:

* Children with mental and motor development retardation
* Patients scheduled emergency surgery
* Patients and parents, who refused to participate in this study

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric patients between 2 months to 18 years undergoing any surgery was included on this study. Pain of these patients' will be evaluated by many pain scales in the postoperative period. These scales include OUCHER, Visiuel Analog Scale, FLACC, Faces Pain Scale revise, Wong Baker Faces Scale, Faces Pain Scale, Numeric rating Scale, Verbal Rating Scale, CHEOPS and also age, blood pressure, respiratuar rate, heart rate will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Artificial Neural Network | 4 months
  the creation of new pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Özcengiz, Principal Investigator — Cukurova University
Locations (1):
- Zehra Hatipoğlu, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Azimi P, Mohammadi HR, Benzel EC, Shahzadi S, Azhari S, Montazeri A. Artificial neural networks in neurosurgery. J Neurol Neurosurg Psychiatry. 2015 Mar;86(3):251-6. doi: 10.1136/jnnp-2014-307807. Epub 2014 Jul 1. PMID 24987050
- See also: Artificial neural networks in neurosurgery — http://www.ncbi.nlm.nih.gov/pubmed/24987050